CLINICAL TRIAL: NCT01625130
Title: Down Regulation of Oxidant Induced Airway Inflammation Through Modulation of NRF2
Brief Title: Effect of Sulforaphane-rich Broccoli Sprout Homogenate on Ozone Induced Inflammation Through Modulation of NRF2
Acronym: BroccOz
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michelle Hernandez, MD, Assistant Professor of Pediatrics, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Crossover | Masking: Triple
Other Study IDs: 11-1296
Record Dates: First submitted 2012-06-19; First posted 2012-06-21 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Healthy
Keywords: sulforaphane; ozone; airway inflammation; broccoli sprouts; NRF2; controls

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- broccoli sprout homogenate (BSH) (Active Comparator): Two hundred grams of BSH is equivalent to approximately 111 grams fresh sprouts (about one 4 oz package). Commercially available Broccosprouts® (Brassica Protection Products LLC) will be homogenized with water.
  Interventions: Dietary Supplement: Broccoli sprout homogenate
- alfalfa sprout homogenate (Placebo Comparator): Two hundred grams of commercially available alfalfa sprouts will be homogenized with water using a ratio of 1:1.2 in a clean blender. The homogenate will then be frozen in aliquots at -20 degrees C.
  Interventions: Dietary Supplement: alfalfa sprout homogenate

INTERVENTIONS:
Dietary Supplement: Broccoli sprout homogenate — Commercially available Broccosprouts® (Brassica Protection Products LLC) will be homogenized with water using a ratio of 1:1.2 in a clean blender. The homogenate will then be frozen in aliquots at -20 degrees C.
  Other Names: Broccosprouts® (Brassica Protection Products LLC)
  Arms: broccoli sprout homogenate (BSH)
Dietary Supplement: alfalfa sprout homogenate — 200 grams of alfalfa sprouts will be homogenized with water using a ratio of 1:1.2 in a clean blender. The homogenate will then be frozen in aliquots at -20 degrees C.
  Arms: alfalfa sprout homogenate

SUMMARY:
Purpose: To determine if modulation of NRF2 with a Sulforaphane enriched supplement modifies responses to O3. Participants: Recruitment of up to 70 healthy volunteers, ages 18-50, for completion of 36 volunteers. Procedures: This is a randomized, placebo controlled 2x2 crossover study of treatment with an NRF2 modifier versus placebo in healthy volunteers which will examine airway inflammation before and 4 hours after a 2 hour 0.4 ppm O3 exposure. Participants will be randomized to received either the NRF2 modifier, SFN oral supplement (i.e. broccoli sprout shake), or placebo (alfalfa shake) for 3 days followed by a 0.4 ppm O3 exposure for 2 hours. At least 2 weeks later subjects will return for a 2nd supplementation treatment (using the alternative supplement to that provided initially) followed by an ozone exposure identical to the initial one.

DETAILED DESCRIPTION:
Potential subjects will be seen for a baseline screening visit at which time informed consent will be obtained, a 12 lead ECG will be performed and spirometry with subsequent sputum induction will be performed. Only subjects meeting the lung function criteria as well as criteria for adequate sputum production will continue in the study. If the sample is considered "borderline" by the study team, the subject maybe invited back to repeat collection of another sputum sample. Subjects will be required to abstain from caffeine for 12 hours prior to all study visits and must not use/ingest non-steroidal anti-inflammatory medications, anti-oxidant vitamins, juices/drinks fortified with extra vitamin supplement and cruciferous vegetables 7 days prior to all visits. Subjects will be provided with a list of cruciferous vegetables.

Qualified volunteers will next be seen for a training visit at which time they will undergo physical exam by a study physician. After baseline spirometry is evaluated, the subject will exercise on a treadmill, and measurements of minute ventilation will be collected. Treadmill speed and/or elevation will be adjusted until the subject's minute ventilation is at the target level of 30-40 L/min. The resulting speed and elevation will be used during the ozone exposure sessions. At the training visit, participants will also undergo nasal epithelial biopsy from one nare, and a buccal swab will be collected for genotyping. Baseline blood samples will also be collected at this time for analyses of markers of inflammation, cytokine assessments, SFN levels and complete blood cell count with differential.

After completion of the training session, the subject will return for 4 sequential days. During the first 3 days, subjects will ingest (observed ingestion) either broccoli sprout homogenate or alfalfa sprout homogenate based on earlier randomization. One hour after the supplement dose on the 3rd day, the volunteer will undergo exposure to 0.4 ppm ozone for a 2 hour period. During exposure, subjects will perform 15 minutes of moderate exercise on a treadmill (minute ventilation = 30-40 L/min), each separated by 15 minutes of seated rest. Heart rate and rhythm will be continuously monitored throughout the exposure. Spirometry and symptom scoring will be performed both prior to and after exposure. One hour after the end of exposure, a nasal epithelial biopsy will be collected from the nare that is contralateral to that used at the prior visit. Four hours after completion of the exposure, blood will be drawn for study endpoints and a sputum induction will be performed. The following day the subject will return for a follow-up visit to include vital signs, symptom scoring, spirometry, sputum induction and venipuncture for blood endpoints.

Subjects will be required to abstain from a list of vegetables for 1 week prior to each study session until the completion of that session. Subjects will also be asked to maintain a food diary for the same time.

After a 2 to 6 weeks washout period, participants will again return for a repeated sequence of 4 days with 3 days of supplement ingestion followed by ozone exposure using the alternate supplement and a 24 hour post exposure follow-up visit. Samples for analyses will be collected at the same time points as those used in the initial sequence.

ELIGIBILITY:
Inclusion Criteria:

1. Normal lung function, defined as (NHanes 2001 set):

   FVC of > 80 % of that predicted for gender, ethnicity, age and height; FEV1 of > 80 % of that predicted for gender, ethnicity, age and height; FEV1/FVC ratio of > .70.
2. Negative pregnancy test for females who are not s/p hysterectomy with oophorectomy;
3. Willing to avoid corticosteroids and non-steroidal anti-inflammatory medications for 1 week prior the baseline screening visit and again for 1 week prior to all remaining visits;
4. Willing to avoid antioxidant vitamins and cruciferous vegetables as well as juices/drinks with added vitamin supplements for 7 days prior the baseline screening visit and throughout initial dosing period and ozone challenge as well as 7 days prior to the start of the 2nd dosing period and subsequent challenge.
5. Willing to abstain from caffeine for 12 hours prior to all visits.Inclusion Criteria:

   -

Exclusion Criteria:

1. Any chronic medical condition considered by the PI as a contraindication to the exposure study including, but not limited to, asthma, significant cardiovascular disease, diabetes, chronic renal or thyroid disease;
2. Use of tricyclics and MAO inhibitors;
3. Pregnancy or nursing a baby;
4. Any current smoking;
5. Viral upper respiratory tract infection within 2 weeks of challenge;
6. Any acute infection requiring antibiotics within 2 weeks of challenge;
7. Abnormal physical findings at the baseline visit:

   Abnormalities on lung auscultation Temperature > 37.8 Systolic BP>150 mm hg or < 85 mm Hg or diastolic BP>90 mm Hg or < 50 Oxygen saturation of < 94%;
8. Subjects must demonstrate the ability to produce an acceptable induced sputum sample during the screening session. If the sample is unsatisfactory, the subject's participation will end at that point;
9. Subjects who have been prescribed daily anti-inflammatory medications or medications for asthma will be excluded. Oral contraceptives are acceptable. Antidepressants and other medications may be permitted if in the opinion of the investigator the medication will not interfere with the study procedures or compromise safety; and if the dosage has been stable for 1 month;
10. Subjects who are unwilling to refrain from strenuous physical activity for 24 hours before and after exposure;
11. Current nutritional disorder such as anorexia, bulimia, irritable bowel syndrome, Crohn's disease etc;
12. Current use of immunosuppressive drugs;
13. History of intolerance of or aversion to broccoli;
14. Inability or unwillingness of a participant to give written informed consent;
15. Receipt of LAIV (Live Attenuated Influenza Vaccine), also known as FluMist®, or other live vaccine within the prior 14 days.
16. Orthopedic injuries or impediments that would preclude treadmill exercise.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-10; Primary Completion 2015-05 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in % neutrophils in induced sputum, comparing the 4 hr post O3 placebo v. SFN treatment periods. | baseline, 4 and 24 hours post exposure
  Induced sputum will be collected and % neutrophils will be measured after each exposure and will be compared to baseline and to each other.

SECONDARY OUTCOMES:
Spirometry (FEV1, FVC, FEF25-75) for assessment of changes in lung function | prior to and after exposures
  Lung function testing will be performed prior to, after and 24 hours post exposure
SFN levels | at baseline (sputum & plasma); immediately before the O3 exposure (plasma), 4 hours & 24 hours post O3 (sputum & plasma).
  Sulforaphane levels will be measured in blood and sputum at predetermined intervals
Cytokine concentration and flow cytometric assessment of surface markers in sputum supernatants | baseline, 4 and 24 hours post exposure
  GM-CSF, IL-1β, IL-6, IL-8, IL-10, IL-12p70, TNF-α, PGE2
mRNA expression of NRF2 and phase II antioxidant enzymes in nasal epithelial cells and in induced sputum macrophages | baseline and 1 hour (nasal epithelial cells only) 4 and 24 hours post exposure (sputum)
  GSTM1, GSTP1, NQO1, and HO1)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle Hernandez, Principal Investigator — University of North Carolina, Chapel Hill School of Medicine
Locations (1):
- UNC Center for Environmental Medicine, Asthma and Lung Biology, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Duran CG, Burbank AJ, Mills KH, Duckworth HR, Aleman MM, Kesic MJ, Peden DB, Pan Y, Zhou H, Hernandez ML. A proof-of-concept clinical study examining the NRF2 activator sulforaphane against neutrophilic airway inflammation. Respir Res. 2016 Jul 22;17(1):89. doi: 10.1186/s12931-016-0406-8. PMID 27450419